CLINICAL TRIAL: NCT01325493
Title: Modulation of μ Opioid Receptor Mediated Analgesia, Tolerance and Hyperalgesia in Children and Adolescents
Brief Title: Low Dose Ketamine Study on Opioid Tolerance and Hyperalgesia
Acronym: KPSF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Julia Finkel (Other)
Responsible Party: Sponsor-Investigator, Julia Finkel, Director of Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4735
Record Dates: First submitted 2011-02-25; First posted 2011-03-29 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Idiopathic Scoliosis; Spondylolisthesis
Keywords: opioid tolerance; hyperalgesia; scoliosis; pupillometry
MeSH Terms: conditions — Spondylolisthesis; Hyperalgesia; Scoliosis | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Normal Saline given 0.5mg/kg intravenous (IV) load followed by an intraoperative continuous infusion at 0.25mg/kg/h and a postoperative infusion at 0.1mg/kg/h
  Interventions: Drug: Normal Saline
- Ketamine (Active Comparator): ketamine 0.5mg/kg intravenous (IV) load followed by an intraoperative continuous infusion at 0.25mg/kg/h and a postoperative infusion at 0.1mg/kg/h
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine 0.5mg/kg intravenous (IV) load followed by an intraoperative continuous infusion at 0.25mg/kg/h and a postoperative infusion at 0.1mg/kg/h
  Other Names: Ketanest, Ketaset, and Ketalar
  Arms: Ketamine
Drug: Normal Saline — Normal saline given 0.5mg/kg intravenous (IV) load followed by an intraoperative continuous infusion at 0.25mg/kg/h and a postoperative infusion at 0.1mg/kg/h
  Other Names: 0.90% NaCl
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to:

1. Establish whether ketamine can decrease opioid consumption and modulate the onset of opioid tolerance and prevent opioid-induced hyperalgesia in pediatric subjects, ages 10 years to 18 years, undergoing posterior spinal fusion and instrumentation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 10 to 18 years of age
2. The subject's American Society of Anesthesiologists physical status is ASA 1, 2 or 3 (see appendix I)
3. The subject is scheduled for elective posterior spinal fusion and instrumentation.
4. The subject's parent/legally authorized guardian has given written informed consent to participate

Exclusion Criteria:

1. The subject has a history or a family (parent or sibling) history of malignant hyperthermia
2. The subject is pregnant or nursing.
3. The subject has known significant renal disorders determined by medical history, physical examination or laboratory tests
4. The subject has a known or suspected allergy to morphine, remifentanil or ketamine
5. The subject is an ASA classification of 4 or greater (See Appendix I)
6. The subject is scheduled for a surgical sub-procedure (i.e. anterior spinal fusion)
7. The subject is unable to self-administer morphine using patient-controlled analgesia (PCA) pump
8. The subject had a recent opioid exposure (within 1 month of surgery)
9. The subject is obese (body mass index >30kg/m2)
10. The subject is planned for elective postoperative ventilation
11. The subject has a known ocular disease not permitting pupillometric examination
12. The subject has used any investigation products in the past 30 days

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pestieau Sophie, MD, Principal Investigator — Children's National Research Institute; Finkel C Julie, MD, Study Director — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Pestieau SR, Finkel JC, Junqueira MM, Cheng Y, Lovejoy JF, Wang J, Quezado Z. Prolonged perioperative infusion of low-dose ketamine does not alter opioid use after pediatric scoliosis surgery. Paediatr Anaesth. 2014 Jun;24(6):582-90. doi: 10.1111/pan.12417. PMID 24809838

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Ketamine was diluted in 50mL of normal saline to a concentration of 10 mg*ml-1, administered by the anestheisologist (blind) via IV using a loading dose of 0.5 mg/kg-1, intra-operatively 0.25 mg/kg/hr-1, post-operatively 0.1 mg/kg/hr-1.
- Saline: Normal saline was administered by the anesthesiologist (blind) via IV using a loading dose of 0.5 mg/kg-1, intra-operatively 0.25 mg/kg/hr-1, post-operatively 0.1 mg/kg/hr-1.
Period: Overall Study
Arm/Group | Ketamine | Saline
Started | 30 | 24
Completed | 29 | 21
Not Completed | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — loss of neuromonitoring signals | 0 | 2
Not completed — Allergy | 1 | 0

BASELINE CHARACTERISTICS:
Population: ASA classifications: ASA Physical Status 1 - A normal healthy patient ASA Physical Status 2 - A patient with mild systemic disease ASA Physical Status 3 - A patient with severe systemic disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Saline | Total
Number analyzed (Participants) | 29 | 21 | 50
Age, Continuous [Median (Full Range); unit: years] | 14 [11 to 18] | 14 [12 to 18] | 14 [11 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 38
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 29 | 21 | 50
American Society of Anesthesiology classification [Number; unit: participants] — ASA classifications: ASA Physical Status 1 - A normal healthy patient ASA Physical Status 2 - A patient with mild systemic disease ASA Physical Status 3 - A patient with severe systemic disease
  participants
    ASA 1 | 13 | 14 | 27
    ASA 2 | 15 | 7 | 22
    ASA 3 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalent Consumption (mg/kg)
Description: Morphine consumption (mg/kg) was measured over time in the Ketamine group and compared to the Control (saline) group. Values are for each 24 hour time period and displayed as hours post surgery.
Time Frame: at 24, 48, 72, 96 hours post operatively
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 29 | 21
mg/kg
  24 hrs after surgery | 1.3 (.3) | 1.36 (.42)
  48 hrs after surgery | 1.28 (.26) | 1.275 (.31)
  72 hrs after surgery | .89 (.55) | .93 (.36)
  96 hrs after surgery | .57 (.44) | .38 (.35)

2. Secondary Outcome: Sedation Score
Description: Sedation scores 0 = completely awake
  1. = sleepy but responds appropriately
  2. = somnolent but arouses to light stimuli
  3. = asleep but responsive to deeper physical stimuli
  4. = asleep and not responsive to any stimuli Values are for each 24 hour time period and displayed as hours post surgery.
Time Frame: 24, 48, 72, 96 hours post operatively
Measure: Mean (Standard Deviation); unit: Sedation Score
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 29 | 21
Sedation Score
  24 hrs after surgery | .73 (.68) | .75 (.73)
  48 hrs after surgery | .62 (.8) | .54 (.85)
  72 hrs after surgery | .38 (.45) | .3 (.84)
  96 hrs after surgery | .24 (.43) | .21 (.39)

3. Secondary Outcome: Pain Score at Rest
Description: Patient volunteered response at rest, 1-10 scale (where a higher score indicates more pain and a lower score indicates less pain). Values are for each 24 hour time period and displayed as hours post surgery.
Time Frame: 24, 48, 72, 96 hours post operatively
Measure: Mean (Standard Deviation); unit: pain score at rest
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 29 | 21
pain score at rest
  24 hrs after surgery | 3.9 (2.1) | 4.55 (2.0)
  48 hrs after surgery | 4.53 (1.69) | 5.2 (2.2)
  72 hrs after surgery | 3.6 (2.3) | 3.48 (2.0)
  96 hrs after surgery | 4.48 (2.1) | 3.8 (1.8)

4. Secondary Outcome: Pain Score During Cough.
Description: Patient volunteered response during a cough, 1-10 scale (where a higher score indicates more pain and a lower score indicates less pain). Values are for each 24 hour time period and displayed as hours post surgery.
Time Frame: 24, 48, 72, 96 hours post operatively
Measure: Mean (Standard Deviation); unit: pain score at cough
Arm/Group | Ketamine | Saline
Number analyzed (Participants) | 29 | 21
pain score at cough
  24 hrs after surgery | 4.5 (2.5) | 5.1 (3.0)
  48 hrs after surgery | 5.4 (2.3) | 5.45 (2.7)
  72 hrs after surgery | 4.4 (2.3) | 3.7 (2.5)
  96 hrs after surgery | 5.15 (2.5) | 4.2 (2)

ADVERSE EVENTS:
Time Frame: the duration of the study (96 hrs) post surgery
Arm/Group | Ketamine | Saline
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/21
Other Adverse Events (participants affected / at risk) | 0/29 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=29) | Saline (N=21)
Allergy (Surgical and medical procedures) | 1 (1) | 0 (0) — Morphine allergy

LIMITATIONS AND CAVEATS:
Patient sex and ethnicity could have led to analytical bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No